CLINICAL TRIAL: NCT02455752
Title: Laparoscopic Extraperitoneal Total Mesorectal Excision (LE-TME): A New Feasible Technical Approach.
Acronym: LE-TME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: West oncologic center, Nantes, France (Unknown); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Principal Investigator, Osama Mohammad Ali ElDamshety, Assisstant Lecturer of surgical oncology, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTME-200315
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Total Mesorectal Excision; Laparoscopic
Keywords: LE-TME; Laparoscopic rectal resection; Retroperitoneal resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reroperitoneal Group (Active Comparator): LE-TME
  Interventions: Procedure: LE-TME

INTERVENTIONS:
Procedure: LE-TME — Retroperitoneal approach for total mesorectal excision

SUMMARY:
The study involves the use of Retroperitoneal plane for TME for rectal anterior resection. Through a pilot prospective study, LR-TME will be assessed as one arm study.

DETAILED DESCRIPTION:
This study is based on our new suggested theory for a retro-peritoneal approach. After successful 2 cases of Laparoscopic extraperitoneal-TME. A pilot study for assessment of the feasibilty of the new approach.

Data will be registered prospectively and the perioperative outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* (Rectum, Anal or sigmoid) Malignancy requiring mesorectal excision and Fit for laparoscopic surgery

Exclusion Criteria:

* contraindication to laparoscopic surgery-unwilling to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of the procedure | 1 day
  Feasibility of the TME by the retroperitoneal approach.

SECONDARY OUTCOMES:
Intraoperative morbidity | 1 day
  Intraoperative morbidity including Urteric injury, Vascular injuries, hypogastric nerve injury, intestinal loop injury.
Postoperative morbidity | Till patient discharge
  Postoperative haematoma, colonic leak and/or necrosis, pelvic abscess, intestinal obstruction
Pathologic report outcome | 7 days
  Lymph node harvest, radial and circumferential margin, complete total mesorectal excison

CONTACTS AND LOCATIONS:
Overall Officials: Osama Eldamshety, PhD, Principal Investigator — 1-Assistant lecturer of surgical oncology, Mansoura university Egypt. 2-Research Fellow, Policlinico Umberto primo, LA SAPIENZA, Roma, Italy.; Frédéric Dumont, M.D., Principal Investigator — 1- Department of Digestive Oncological surgery, West oncologic center, Nantes, France 2- Department of digestive Oncological surgery, Gustave Roussy Cancer Campus, Villejuif, France
Locations (1):
- Oncology center of mansoura university, Al Mansurah, Eldakahlia, Egypt